CLINICAL TRIAL: NCT03473535
Title: The BEACON Study: Protocol for a Pilot Randomized Controlled Trial of Smartphone-assisted Problem Solving Therapy in Men Who Present With Intentional Self-harm to Emergency Departments in Ontario
Brief Title: BEACON Suicide Prevention in Men Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ottawa (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Vice-Chair, Department of Psychiatry, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-0790-B
Record Dates: First submitted 2018-02-27; First posted 2018-03-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Intentional Self-Harm; Suicide
Keywords: self-harm; problem-solving therapy; emergency department; e-therapy; suicide prevention
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Emergencies; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PST Alone (Active Comparator): Participants will receive six sessions of face-to-face PST.
  Interventions: Behavioral: Problem-Solving Therapy
- Blended-Therapy (Experimental): Participants with receive six sessions of face-to-face PST supplemented by the BEACON platform.
  Interventions: Combination Product: BEACON + Problem Solving Therapy

INTERVENTIONS:
Combination Product: BEACON + Problem Solving Therapy — Six sessions of face-to-face PST delivered by a trained Research Therapist and access to the BEACON Suicide Prevention smartphone application.
  Arms: Blended-Therapy
Behavioral: Problem-Solving Therapy — Six sessions of face-to-face PST delivered by a trained Research Therapist.
  Arms: PST Alone

SUMMARY:
The purpose of this study is to evaluate the use of problem-solving therapy (PST), supplemented by a smartphone application, in the treatment of men who present to the Emergency Departments in Ontario. A total of 100 men in 5 Emergency Departments will be enrolled and randomized to receive either face-to-face PST or face-to-face PST supplemented by the BEACON Suicide Prevention smartphone application. Face-to-face therapy may be provided via videoconference to accommodate patient preference and ongoing pandemic restrictions. Participants will complete six sessions of PST and outcomes will be measured at baseline, 6 weeks, two post-therapy follow-up time points (3 and 6 months). Participants will also be asked to complete a qualitative interview about their participation in the study and their experience with the smartphone application.

DETAILED DESCRIPTION:
Self-harm is defined as intentional self-poisoning or self-injury, whether or not there is evidence that the act was intended to result in death. In the past, the term used was 'attempted suicide.' However, peoples' motives for harming themselves are highly variable, a person may have more than one motive and motivation is hard to assess. In line with usual public policy in health and social care, we use the term 'self-harm' to describe a behaviour - avoiding the word 'deliberate' because many service users or consumers dislike its connotations.

In Ontario, the number of people who present to hospital emergency departments (ED) with self-harm is difficult to accurately assess and often underreported. Data from CIHI results in an estimated 8,250 ED visits annually (as of 2014) in Ontario. However, using data from Ottawa, Ontario EDs the rate of presentation appears to be more than double at 1,600 presentations annually. Therefore, it is possible that the provincial rate may exceed 16,000 unique presentations. The most common form of self-harm seen in emergency departments (around 80% of episodes) is the intentional consumption of an excess of a medicinal or toxic product, whether or not there is evidence that the act was intended to result in death. Injuries, most commonly self-cutting, form 15-20% of episodes.

Two-thirds of people attending emergency departments because of self-harm are under 35 years of age. They are high users of health and social care services. Self-harm also has a strong association with suicide: 7 patients per 1000 (approximately 1.6%) die by suicide in the year after attending emergency departments with a non-fatal episode, with the incidence rate nearly double in men compared to women, representing a risk nearly 50 times greater than the general population. All-cause mortality is also higher for individuals who self-harm, with significantly more deaths from natural causes and accidents than in the general population. As such, self-harm is associated with a 40-year reduction in average life expectancy. Whilst only four of ten people who present with self-harm are men, they account for nearly two-thirds of suicides after an episode and are far more likely than women to die a premature death from other causes. The rates are even more pronounced in indigenous communities, with suicide rates of 126 per 100,000 young men (15-24) compared to a rate of 24 per 100,000 in non-Indigenous men of the same age.

Approximately 10% of those who present in an Emergency Department following self-harm will engage in repeat self-harm in the following month and up to 27% after six months. Recurrent self-harm is associated with significant distress and many unresolved interpersonal problems. It is likely that any reduction in repetition of self-harm will be mirrored by a fall in subsequent suicides. The Canadian Association for Suicide Prevention blueprint for a National Suicide Prevention Strategy (CASP) has identified those who have presented to the hospital with non-fatal self-harm as a high-risk target group to reduce suicide.

People attending emergency departments after self-harm receive a variable standard of care in Ontario, and there is no standard protocol for therapy. Many are not assessed for psychological needs, and the little psychological therapy available is not usually covered by Ontario Health Insurance (OHIP). Local data from hospitals in Ottawa show that only 4 out of 10 men who present with intentional self-harm are seen by a mental health professional. Few are offered an evidence-based treatment aimed at reducing their risk of suicide or repeated self-harm. Assessment of suicide risk is currently a Required Operating Practice for Canadian Hospital accreditation; however, individuals identified as at-risk for suicide rarely receive recommended care.

Specialist services, when offered, typically include intensive and lengthy treatments such as dialectical behaviour therapy or mindfulness-based therapy. The evidence for the effectiveness of these specialist therapies comes almost entirely from studies in women. Problem-solving therapy (PST) has been identified as a promising intervention in the treatment of self-harm. PST seeks to improve an individual's ability to cope better with both minor (e.g., chronic daily problems) and major (e.g., traumatic events) life stresses to increase mental and physical health. The major goals of PST are to help individuals adopt a positive worldview and way of approaching their problems and increase problem-solving skills in order to better cope with life stressors.

The investigators have received funding for a multi-site individual randomized control trial (RCT) from the Ontario Strategy for Patient Oriented Research (SPOR), Support for People and Patient Oriented Research and Trials (SUPPORT), Unit funded by Canadian Institutes for Health Research, (CIHR) and the Ontario Ministries of Health and Research and Innovation (MRI) studying the feasibility and effectiveness of PST with the use of the BEACON smartphone application compared to PST alone in men who present to Emergency Departments with intentional self-harm. The rationale for focusing on men is that they are less likely to seek care but represent nearly two-thirds of those who die by suicide after an index episode of self-harm, and previous trials have found that providing generic treatments to everyone does not work. The intervention will build on previous work by trying to extend the range and intensity of therapy. The investigators will do this by supplementing PST with a sophisticated smartphone application (BEACON) that has already demonstrated its effectiveness in men with substance abuse disorders. For the purpose of this study, the smartphone application has been re-designed for the treatment of self-harm.

Participants that consent to take part in this study will be assigned randomly to one of two groups: a "control" group and a study intervention group. Both groups receive six free one-on-one sessions of PST over a period of eight weeks. If placed in the control group, the participant will only receive problem-solving therapy and treatment as usual. The intervention group will receive problem-solving therapy, delivered in the same manner, but will be provided access to a smartphone application (BEACON) designed to support the therapy. Eligible participants will consist of men 18 years of age or older who have presented via the Emergency Department of a recruiting site for self-harm and agree to participate in the study. Participants will be asked to complete a series of outcome measures assessing suicidal thoughts and behaviour, problem-solving, mental health and substance use, quality of life and health care service use. These outcomes will be completed at baseline, 6 weeks, 3 months and 6 months. Participants will also be asked to participate in a qualitative interview at the end of the study to gather information on their experience of being in the study, barriers or facilitators to participation and the use of the smartphone application. PST sessions will be delivered by a trained Research Therapist. PST Sessions and other study visits may take place over videoconference, using an approved platform.

Categorical participant characteristics, such as gender identity, marital status and education level will be reported using frequencies and percentages. Continuous characteristics, such as age, will be reported using mean ±SD for any continuous variables that are normally distributed, and as a median score. For non-normally distributed variables the 25th and 75th percentiles will be used. Non-normally distributed variables will also be dichotomized and analyzed as categorical data. Changes in participants' scores from their baseline visit to follow-up at six months will be analyzed by use of repeated measures ANOVA with a generalized linear mixed modelling (GLMM) to account for missing variables. Multivariate linear regression analyses will be performed to determine which participant characteristics moderate primary and secondary treatment outcomes. Additional subgroup analyses will be carried out to determine the impact of smartphone-assisted PST for the following subgroups: first-time presentations of self-harm compared to repeaters; Francophone versus Anglophone; men with substance abuse disorders versus no substance abuse disorder; and rural versus urban residence.

Randomization for this study will occur with 2:1 (67:33) allocation in favour of the blended therapy model. Given the small sample size, there will be no stratification across sites to ensure an equitable allocation to the conditions. A web randomization system hosted by the Ottawa Methods Centre (OMC) will be used. Participants will be randomized by each site coordinator using the web system as they are enrolled. There is no blinding in this study as all patients who consent to participate in this study will receive at least PST therapy. It would not be practical or possible to blind the receipt of the mobile application as both the participant and therapist will be using the platform.

The primary outcome measure is the Beck Scale for Suicide Ideation (BSS), a 24-item self-report questionnaire for detecting and measuring the current intensity of a subject's thoughts, feelings and suicidal behaviours. Secondary outcome measures include: the 9-Item Patient Health Questionnaire (PHQ-9), the Generalized Anxiety Disorder Questionnaire (GAD-7), the Primary Care Post-Traumatic Stress Disorder (PC-PTSD-5) screening tool, the EuroQol 5 Dimensions (EQ-5D-5L) questionnaire, the Experienced Meaning in Life (EMIL) scale, the Multidimensional Scale of Perceived Social Support (MSPSS), the Alcohol Use Disorder Identification Test (AUDIT), the Drug Abuse Screening Test (DAST-10), and two sub-scales from the Conformity to Masculine Norms Scale (CMNI). In order to assess the impact of the intervention on a participant's social problem-solving skills, the Social Problem Solving Inventory-Revised Short Form (SPSI-R:S) will be used, and health service use will be captured using the Questionnaire on Healthcare Consumption and Productivity losses for patients with a Psychiatric Disorder (TiC-P). We will also use routinely collected administrative data obtained from the Institute for Clinical Evaluative Sciences (ICES). The ICES data collected will characterize a participant's previous hospitalizations for self-harm, previous presentations to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to the hospital for any reason, outpatient appointments for any reason, and primary care visits.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as Male.
* 18 years of age or older.
* Has presented via the Emergency Department with self-harm in the preceding 4 weeks
* Able to read and understand English, French or read or understand Oji Cree.
* Willing to attend six problem-solving therapy sessions for a period of up to eight weeks.
* Willing to use a smartphone application to facilitate the treatment of self-harm.
* Willing to return to the hospital for follow-up appointments.
* Willing and able to provide informed consent.
* Willing to use e-mail for study activities.

Exclusion Criteria:

* Identifies as female.
* Has presented to the Emergency Department for a reason other than self-harm.
* In the opinion of the investigator is unlikely to commit to a six-month long study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who identify as male will be eligible for participation in the trial.
Enrollment: 100 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-09-23 (Estimated)

PRIMARY OUTCOMES:
Change in Measure of Suicidality - 24-Item Beck Scale for Suicidal Ideation (BSS) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported measurement of the current intensity of a participant's attitudes, behaviours, and plans to die by suicide during the past week. It consists of 5 screening items, and 19 follow-up items. Each item is scored from 0 (moderate to strong) to 2 (none), yielding a total score ranging from 0 to 48, with higher scores indicating a higher risk of suicidality. Generally, scores above 24 are considered to be a clinical cutoff implying that the respondent is at significant risk for suicide.

SECONDARY OUTCOMES:
Change in Severity of Depression Symptoms - 9-Item Patient Health Questionnaire (PHQ-9) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported measurement of the severity of depression symptoms experienced within the last two weeks. The survey consists of 9 items. Participants are asked to rate each symptom of depression on a Likert scale, providing a score between 0 (not at all) and 3 (nearly every day). This yields a total score ranging from 0 (minimal depression) to 27 (severe depression). Higher scores thus indicate a greater severity of depressive symptoms, and are interpreted in the following manner: a score of 0-4 indicates minimal depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, a score of 15-19 indicates moderately severe depression, and a score of 20-27 indicates severe depression.
Change in Severity of Anxiety Symptoms - 7-Item General Anxiety Disorder Questionnaire (GAD-7) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported measurement of the severity of anxiety symptoms experienced within the last two weeks. It consists of 7 scored items and one follow-up question. Each of the 7 scored items generates a value from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0 to 21, with higher scores indicating more severe symptoms of anxiety. These scores are interpreted in the following manner: a score of 0-4 indicates little or no anxiety, a score of 5-9 indicates mild anxiety, a score of 10-14 indicates moderate anxiety, and a score of 15-21 indicates severe anxiety. Generally, a score of 10 or above is considered to be a clinical cutoff implying that the respondent may be suffering from a general anxiety disorder.
Change in Post-Traumatic Stress Disorder Symptoms - 5-Item Primary Care Post-Traumatic Stress Disorder Screening Tool for DSM-5 (PC-PTSD-5) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing the presence of PTSD-related symptoms. The questionnaire consists of five items requiring a 'yes' or 'no' response. The result of the questionnaire is either 'positive' or 'negative' based on the number of 'yes' responses indicated. The authors suggest that the results of the PC-PTSD-5 survey should be considered 'positive' if three or more yes responses are indicated. A 'positive' result on this questionnaire suggests that the respondent has probable PTSD.
Change in Health-Related Quality of Life - 5-Item EuroQol 5 Dimensions Questionnaire (EQ-5D-5L) | Baseline; Session 6; 3 months; 6 months Post-Enrollment
  Self-reported questionnaire assessing 5 health-related dimensions relevant to quality of life. These dimensions consist of mobility, self-care, ability to participate in one's usual activities, pain or discomfort, and anxiety or depression. Each dimension consists of 5 items, which are ranked by means of a Likert scale from 1 to 5. A score of 1 in a given dimension indicates no problems for that dimension of health, a score of 2 indicates slight problems for dimension, a score of 3 indicates moderate problems for that dimension, a score of 4 indicates severe problems for that dimension, and a score of 5 indicates extreme problems for that dimension. Respondent decisions result in a 1 digit number expressing the level selected for that dimension. The digits for these five dimensions are combined, resulting in a five digit number, and indicating one of 3,125 possible health states. This five digit number has no arithmetic properties, and is not used as a cardinal score.
Change in Health-Related Quality of Life - 5-Item EuroQol 5 Dimensions Questionnaire (EQ-5D-5L): Visual Analogue Scale (VAS) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing health-related quality of life, including mobility, self-care, ability to participate in one's usual activities, pain or discomfort, and anxiety or depression. It consists of 5 items, which are ranked by means of a Likert scale from 1 to 5. Respondents fall into one of 3,125 different health states depending on their responses to the questionnaire. The measure also includes a Visual Analogue Scale (VAS) which asks participants to evaluate their overall health on a scale from 0-100. Higher scores on the VAS scale indicate a better state of general health, with a score of 100 suggesting the "best imaginable health state" and a score of 0 suggesting the "worst imaginable health state."
Change in Meaning in Life - 40-Item Experienced Meaning in Life Questionnaire (EMIL): Four sub-scales (Creative, Experiential, Attitudinal, Ultimate) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing a participant's perceived meaning in life. The full EMIL survey consists of four 10-item sub-scales rated on a Likert scale, with each item generating a number between 1 (strongly disagree) to 5 (strongly agree). This produces a total score ranging from 40 to 200. Higher scores reflect greater perceived meaning in life.
Change in Perceived Social Supports - 12-Item Multidimensional Scale of Perceived Social Supports (MSPSS) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing a respondents perceived level of social supports available. It consists of 12 items rated on a seven-point Likert scale, generating scores between 1 (very strongly disagree) and 7 (very strongly agree). Items are arranged into three subscales (Significant Other, Family, and Friends) consisting of four items each. Mean scores are generated for each sub-scale by adding the values together and dividing by four. A total value is generated by adding together all values and dividing by 12, resulting in a mean scale score between 1 and 7, with higher scores indicating a higher level of perceived social support. These scores can be interpreted in the following manner: a score between 1 and 2.9 could be considered low support, a score between 3 and 5 can be considered moderate support, and a score from 5.1 to 7 can be considered high support.
Change in Alcohol Misuse - 3-Item Alcohol Use Disorder Identification Test (AUDIT-C) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing alcohol consumption, drinking behaviour, adverse reactions, and alcohol-related problems. Two versions of the AUDIT questionnaire will be used in this study. The 3 item version (AUDIT-C) will be employed as a screening questionnaire, and the full 10 item version employed as a follow-up questionnaire. Each of the 10 items generates a score between 0 (never) and 4 (daily or almost daily), with a total score generated by summing the values. The AUDIT-C survey generates a score between 0 and 12, with higher scores indicating a greater risk of alcoholism. Given that higher scores act as an indicator that respondents have problems with alcohol, participants with a score of above 4 on the AUDIT-C will be asked to complete the full questionnaire.
Change in Alcohol Misuse - 10-Item Alcohol Use Disorder Identification Test (AUDIT) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing alcohol consumption, drinking behaviour, adverse reactions, and alcohol-related problems. Two versions of the AUDIT questionnaire will be used in this study. The 3 item version (AUDIT-C) will be employed as a screening questionnaire, and the full 10 item version employed as a follow-up questionnaire. Each of the 10 items generates a score between 0 (never) and 4 (daily or almost daily), with a total score generated by summing the values. Scoring on the full AUDIT questionnaire generates a total ranging between 0 and 40, with higher scores acting as an indicator that respondents have problems with alcohol. AUDIT scores of 8 or above are recommended as indicators of hazardous and harmful alcohol use. A score of between 8 and 15 represents a medium level of alcohol problems, and a score of 16 or above represents a high level of alcohol problems.
Change in Drug Misuse - 10-Item Drug-Abuse Screening Test (DAST-10) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing drug abuse within the last 12 months. It consists of 10 items requiring a 'yes' or 'no' response. Each response indicating a possible drug-use problem is awarded one point. Total scores range between 0 and 10, with higher scores acting as an indicator that the respondent has a substance abuse problem. A score of 0 suggests no problems, a score of 1-2 suggests a low level of drug abuse problems, a score of 3-5 suggests a moderate level of drug abuse problems, a score of 6-8 suggests a substantial level of drug abuse problems, and a score of 9-10 suggests a severe level of drug abuse problems.
Adherence to Masculine Gender Roles - 94-Item Conformity to Masculine Norms Scale (CMNI): Emotional Control Sub-Scale | Baseline Visit
  Self-reported questionnaire assessing a participant's personal conformity with masculine gender norms. The full CMNI questionnaire consists of 94 items rated on a four-point Likert scale, generating scores between 1 (strongly disagree) and 4 (strongly agree). This produces a total score ranging between 94 and 376. For the purposes of this study, the investigators will only be using the Emotional Control (CMNI-EC) and Self-Reliance (CMNI-SR) sub-scales in order to reduce the burden on participants and study staff. The emotional control sub-scale consists of 12 questions, and generates a score between 12 and 48, with higher scores indicating greater conformity to masculine norms as regards emotion.
Adherence to Masculine Gender Roles - 94-Item Conformity to Masculine Norms Scale (CMNI): Self-Reliance Sub-Scale | Baseline Visit
  Self-reported questionnaire assessing a participant's personal conformity with masculine gender norms. The full CMNI questionnaire consists of 94 items rated on a four-point Likert scale, generating scores between 1 (strongly disagree) and 4 (strongly agree). This produces a total score ranging between 94 and 376. For the purposes of this study, the investigators will only be using the Emotional Control (CMNI-EC) and Self-Reliance (CMNI-SR) sub-scales in order to reduce the burden on participants and study staff. The self-reliance sub-scale consists of 12 questions, and generates a score between 12 and 48, with higher scores indicating greater conformity to masculine norms as regards self-reliance.
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Previous Hospitalizations for Self-Harm | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits. This particular outcome item refers to "previous hospitalizations for self-harm". The incidence of previous hospitalizations for self-harm will be measured using the ICD-10-CM codes T360-T50992, T510-T6592, T71112-T71232, and X71-X83.
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Presentation to Hospital for Self-Harm | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits.
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Presentations to the Hospital for Any Reason Other Than Self-Harm | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits. A questionnaire has also been created by the research team to capture data not available in ICES. Specifically, elements from the Client Service Receipt Inventory (CSRI) and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) have been integrated for the purposes of gathering the above-listed data. This particular outcome item refers to "Presentations to the Hospital for any Reason Other Than Self-Harm."
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Admission to the Hospital for Any Reason. | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits. A questionnaire has also been created by the research team to capture data not available in ICES. Specifically, elements from the Client Service Receipt Inventory (CSRI) and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) have been integrated for the purposes of gathering the above-listed data. This particular outcome item refers to "Admission to the Hospital for Any Reason."
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Outpatient Appointment for Any Reason. | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits. A questionnaire has also been created by the research team to capture data not available in ICES. Specifically, elements from the Client Service Receipt Inventory (CSRI) and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) have been integrated for the purposes of gathering the above-listed data. This particular outcome item refers to "Outpatient Appointment for Any Reason."
Health Service Use - Data from the Institute for Clinical Evaluative Sciences (ICES): Primary Care Visits. | 6 months Post-Enrollment.
  Health service use will be captured using routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES). Data to be collected includes: previous hospitalizations for self-harm, presentation to hospital for self-harm, presentations to hospital for any reason other than self-harm, admission to hospital for any reason, outpatient appointment for any reason, and primary care visits. A questionnaire has also been created by the research team to capture data not available in ICES. Specifically, elements from the Client Service Receipt Inventory (CSRI) and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) have been integrated for the purposes of gathering the above-listed data. This particular outcome item refers to "Primary Care Visits."
Problem-Solving Skills - 25-Item Social Problem Solving Inventory - Revised Short Form (SPSI-R:S) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Self-reported questionnaire assessing the impact of the intervention (smartphone-assisted Problem Solving Therapy) on a participants social problem solving skills. The questionnaire consists of 25 items and 5 scales (positive problem orientation, rational problem-solving style, negative problem orientation, impulsivity/carelessness style, and avoidance style). Participants are asked to choose one of five possible responses for each item, generating a score between 0 and 4. This yields a total score ranging between 0 and 100, with higher scores indicating an individual with more effective problem-solving skills.
Health Service Use - Questionnaire on Healthcare Consumption and Productivity losses for patients with a Psychiatric Disorder (TiC-P) | Baseline; Session 6; 3 months; 6 months Post-Enrollment.
  Health service use (healthcare consumption) and work productivity will be captured using the TiC-P. The TiC-P is a 29-item self-report questionnaire taking less than 10 minutes to complete. Some items have been removed or modified from the original TiC-P including optional items as noted by the developers, items captured elsewhere in a more reliable manner (such as current medications or demographics), or items adapted to better describe services in Ontario healthcare system.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatcher, PhD, Principal Investigator — University of Ottawa; Marnin Heisel, PhD, Principal Investigator — Western University, Canada
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klonsky ED. Non-suicidal self-injury in United States adults: prevalence, sociodemographics, topography and functions. Psychol Med. 2011 Sep;41(9):1981-6. doi: 10.1017/S0033291710002497. Epub 2011 Jan 5. PMID 21208494
- [Background] Gunnell D, Bennewith O, Peters TJ, House A, Hawton K. The epidemiology and management of self-harm amongst adults in England. J Public Health (Oxf). 2005 Mar;27(1):67-73. doi: 10.1093/pubmed/fdh192. Epub 2004 Nov 25. PMID 15564277
- [Background] Hawton K, Bergen H, Casey D, Simkin S, Palmer B, Cooper J, Kapur N, Horrocks J, House A, Lilley R, Noble R, Owens D. Self-harm in England: a tale of three cities. Multicentre study of self-harm. Soc Psychiatry Psychiatr Epidemiol. 2007 Jul;42(7):513-21. doi: 10.1007/s00127-007-0199-7. Epub 2007 May 21. PMID 17516016
- [Background] Carroll R, Metcalfe C, Gunnell D. Hospital presenting self-harm and risk of fatal and non-fatal repetition: systematic review and meta-analysis. PLoS One. 2014 Feb 28;9(2):e89944. doi: 10.1371/journal.pone.0089944. eCollection 2014. PMID 24587141
- [Background] Finkelstein Y, Macdonald EM, Hollands S, Sivilotti ML, Hutson JR, Mamdani MM, Koren G, Juurlink DN; Canadian Drug Safety and Effectiveness Research Network (CDSERN). Risk of Suicide Following Deliberate Self-poisoning. JAMA Psychiatry. 2015 Jun;72(6):570-5. doi: 10.1001/jamapsychiatry.2014.3188. PMID 25830811
- [Background] Eynan R, Shah R, Heisel MJ, Eden D, Jhirad R, Links PS. The Feasibility and Clinical Utility of Conducting a Confidential Inquiry Into Suicide in Southwestern Ontario. Crisis. 2018 Jul;39(4):283-293. doi: 10.1027/0227-5910/a000500. Epub 2017 Dec 19. PMID 29256267
- [Background] Owens D, House A. General hospital services for deliberate self-harm. Haphazard clinical provision, little research, no central strategy. J R Coll Physicians Lond. 1994 Jul-Aug;28(4):370-1. No abstract available. PMID 7965981
- [Background] Da Cruz D, Pearson A, Saini P, Miles C, While D, Swinson N, Williams A, Shaw J, Appleby L, Kapur N. Emergency department contact prior to suicide in mental health patients. Emerg Med J. 2011 Jun;28(6):467-71. doi: 10.1136/emj.2009.081869. Epub 2010 Jul 26. PMID 20660941
- [Background] Hawton K, Harriss L, Zahl D. Deaths from all causes in a long-term follow-up study of 11,583 deliberate self-harm patients. Psychol Med. 2006 Mar;36(3):397-405. doi: 10.1017/S0033291705006914. Epub 2006 Jan 10. PMID 16403244
- [Background] Comtois KA, Russo J, Snowden M, Srebnik D, Ries R, Roy-Byrne P. Factors associated with high use of public mental health services by persons with borderline personality disorder. Psychiatr Serv. 2003 Aug;54(8):1149-54. doi: 10.1176/appi.ps.54.8.1149. PMID 12883144
- [Background] Owens D, Horrocks J, House A. Fatal and non-fatal repetition of self-harm. Systematic review. Br J Psychiatry. 2002 Sep;181:193-9. doi: 10.1192/bjp.181.3.193. PMID 12204922
- [Background] Milnes D, Owens D, Blenkiron P. Problems reported by self-harm patients: perception, hopelessness, and suicidal intent. J Psychosom Res. 2002 Sep;53(3):819-22. doi: 10.1016/s0022-3999(02)00327-6. PMID 12217457
- [Background] Ness J, Hawton K, Bergen H, Cooper J, Steeg S, Kapur N, Clarke M, Waters K. Alcohol use and misuse, self-harm and subsequent mortality: an epidemiological and longitudinal study from the multicentre study of self-harm in England. Emerg Med J. 2015 Oct;32(10):793-9. doi: 10.1136/emermed-2013-202753. Epub 2015 Jan 6. PMID 25564479
- [Background] Hawton K, Witt KG, Taylor Salisbury TL, Arensman E, Gunnell D, Hazell P, Townsend E, van Heeringen K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2016 May 12;2016(5):CD012189. doi: 10.1002/14651858.CD012189. PMID 27168519
- [Background] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- [Background] Haw C, Hawton K, Casey D, Bale E, Shepherd A. Alcohol dependence, excessive drinking and deliberate self-harm: trends and patterns in Oxford, 1989-2002. Soc Psychiatry Psychiatr Epidemiol. 2005 Dec;40(12):964-71. doi: 10.1007/s00127-005-0981-3. Epub 2005 Dec 9. PMID 16341616
- [Background] Krieger T, Meyer B, Sude K, Urech A, Maercker A, Berger T. Evaluating an e-mental health program ("deprexis") as adjunctive treatment tool in psychotherapy for depression: design of a pragmatic randomized controlled trial. BMC Psychiatry. 2014 Oct 8;14:285. doi: 10.1186/s12888-014-0285-9. PMID 25298158
- [Background] Kooistra LC, Wiersma JE, Ruwaard J, van Oppen P, Smit F, Lokkerbol J, Cuijpers P, Riper H. Blended vs. face-to-face cognitive behavioural treatment for major depression in specialized mental health care: study protocol of a randomized controlled cost-effectiveness trial. BMC Psychiatry. 2014 Oct 18;14:290. doi: 10.1186/s12888-014-0290-z. PMID 25326035
- [Background] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181
- [Background] Reid SC, Kauer SD, Hearps SJ, Crooke AH, Khor AS, Sanci LA, Patton GC. A mobile phone application for the assessment and management of youth mental health problems in primary care: a randomised controlled trial. BMC Fam Pract. 2011 Nov 29;12:131. doi: 10.1186/1471-2296-12-131. PMID 22123031
- [Background] Proudfoot J, Parker G, Hadzi Pavlovic D, Manicavasagar V, Adler E, Whitton A. Community attitudes to the appropriation of mobile phones for monitoring and managing depression, anxiety, and stress. J Med Internet Res. 2010 Dec 19;12(5):e64. doi: 10.2196/jmir.1475. PMID 21169174
- [Background] Cooper J, Steeg S, Bennewith O, Lowe M, Gunnell D, House A, Hawton K, Kapur N. Are hospital services for self-harm getting better? An observational study examining management, service provision and temporal trends in England. BMJ Open. 2013 Nov 19;3(11):e003444. doi: 10.1136/bmjopen-2013-003444. PMID 24253029
- [Background] Olfson M, Marcus SC, Bridge JA. Emergency treatment of deliberate self-harm. Arch Gen Psychiatry. 2012 Jan;69(1):80-8. doi: 10.1001/archgenpsychiatry.2011.108. Epub 2011 Sep 5. PMID 21893643
- [Background] Schoen C, Osborn R, Squires D, Doty M, Rasmussen P, Pierson R, Applebaum S. A survey of primary care doctors in ten countries shows progress in use of health information technology, less in other areas. Health Aff (Millwood). 2012 Dec;31(12):2805-16. doi: 10.1377/hlthaff.2012.0884. Epub 2012 Nov 15. PMID 23154997
- [Background] Tyrer P, Thompson S, Schmidt U, Jones V, Knapp M, Davidson K, Catalan J, Airlie J, Baxter S, Byford S, Byrne G, Cameron S, Caplan R, Cooper S, Ferguson B, Freeman C, Frost S, Godley J, Greenshields J, Henderson J, Holden N, Keech P, Kim L, Logan K, Manley C, MacLeod A, Murphy R, Patience L, Ramsay L, De Munroz S, Scott J, Seivewright H, Sivakumar K, Tata P, Thornton S, Ukoumunne OC, Wessely S. Randomized controlled trial of brief cognitive behaviour therapy versus treatment as usual in recurrent deliberate self-harm: the POPMACT study. Psychol Med. 2003 Aug;33(6):969-76. doi: 10.1017/s0033291703008171. PMID 12946081
- [Background] Hatcher S, Sharon C, Parag V, Collins N. Problem-solving therapy for people who present to hospital with self-harm: Zelen randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):310-6. doi: 10.1192/bjp.bp.110.090126. Epub 2011 Aug 4. PMID 21816868
- [Background] Akbari A, Mayhew A, Al-Alawi MA, Grimshaw J, Winkens R, Glidewell E, Pritchard C, Thomas R, Fraser C. Interventions to improve outpatient referrals from primary care to secondary care. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD005471. doi: 10.1002/14651858.CD005471.pub2. PMID 18843691
- [Background] Cochrane-Brink KA, Lofchy JS, Sakinofsky I. Clinical rating scales in suicide risk assessment. Gen Hosp Psychiatry. 2000 Nov-Dec;22(6):445-51. doi: 10.1016/s0163-8343(00)00106-7. PMID 11072061
- [Background] Steer RA, Rissmiller DJ, Ranieri WF, Beck AT. Dimensions of suicidal ideation in psychiatric inpatients. Behav Res Ther. 1993 Feb;31(2):229-36. doi: 10.1016/0005-7967(93)90090-h. PMID 8442750
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Carey KB, Carey MP, Chandra PS. Psychometric evaluation of the alcohol use disorders identification test and short drug abuse screening test with psychiatric patients in India. J Clin Psychiatry. 2003 Jul;64(7):767-74. doi: 10.4088/jcp.v64n0705. PMID 12934976
- [Background] Yudko E, Lozhkina O, Fouts A. A comprehensive review of the psychometric properties of the Drug Abuse Screening Test. J Subst Abuse Treat. 2007 Mar;32(2):189-98. doi: 10.1016/j.jsat.2006.08.002. Epub 2006 Nov 21. PMID 17306727
- [Background] Eisler RM, Skidmore JR. Masculine gender role stress. Scale development and component factors in the appraisal of stressful situations. Behav Modif. 1987 Apr;11(2):123-36. doi: 10.1177/01454455870112001. No abstract available. PMID 3508379
- [Background] Stack S. Media coverage as a risk factor in suicide. J Epidemiol Community Health. 2003 Apr;57(4):238-40. doi: 10.1136/jech.57.4.238. PMID 12646535
- [Background] Cheng AT, Hawton K, Lee CT, Chen TH. The influence of media reporting of the suicide of a celebrity on suicide rates: a population-based study. Int J Epidemiol. 2007 Dec;36(6):1229-34. doi: 10.1093/ije/dym196. Epub 2007 Sep 28. PMID 17905808
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Self-Injury Hospitalizations Details for Ontario [Internet]. Ottawa (ON): The Canadian Institute for Health Information. c2018 - [cited 2017 Feb 20] Available from: https://yourhealthsystem.cihi.ca/hsp/indepth?lang=en#/indicator/042/2/C5001/
- [Background] Health Indicators 2013 [Internet]. Ottawa (ON): The Canadian Institute for Health Information. c2013 - [cited 2017 Feb 20] Available from: https://secure.cihi.ca/free_products/HI2013_EN.pdf
- [Background] Heisel MJ, Duberstein PR. Working sensitively and effectively to reduce suicide risk among older adults. In: Kleespies PM, editor. The Oxford handbook of behavioural emergencies and crises. Oxford: Oxford University Press; 2016. P. 335-359.
- [Background] Bergmans Y, Bolton MJ, Hill A, editors. The CASP blueprint for a Canadian national suicide prevention strategy [Internet]. Winnipeg, MB: Canadian Association for Suicide Prevention; 2009 [cited 2017 Feb 20]. Available: https://suicideprevention.ca/wp-content/uploads/2016/09/SuicidePreventionBlueprint0909.pdf
- [Background] Ostamo A, Lonnqvist J. Excess mortality of suicide attempters. Soc Psychiatry Psychiatr Epidemiol. 2001 Jan;36(1):29-35. doi: 10.1007/s001270050287. PMID 11320805
- [Background] Statistics Canada. Canadian coroner and medical examiner database: Annual report (82-214-X) [Internet]. Ottawa: Public Health Agency of Canada; c2012 [cited 2017 May 12] Available from: www.statcan.gc.ca/pub/82-214-x/82-214-x2012001-eng.pdf
- [Background] Accurate: Health Canada. Acting on what we know: Preventing youth suicide in First Nations. [Internet]. Ottawa: Government of Canada; c2010 [cited 2017 December 01] Available from: http://www.hc-sc.gc.ca/fniah-spnia/pubs/promotion/_suicide/prev_youth-jeunes/index-eng.php#tphp
- [Background] Public Health Agency for Northern Ireland. Northern Ireland registry of self-harm western area: Six year summary report 2007-2012 [Internet]. Belfast: Public Health Agency; c2015 [cited February 20 2017] Available from: http://www.publichealth.hscni.net/sites/default/files/Western%20Trust%206-Year%20Report_0.pdf
- [Background] ICD-10-CM: International classification of diseases, 10th revision, clinical modification [Internet]. Atlanta (GA): Center for Disease Control National Center for Health Statistics. C2016 - [cited 2017 May 11] Available from: https:www.cdc.gov/nchs/icd/icd10cm.htm
- [Background] Schull M, Vermeulen T, Stukel T, Fisher E. Follow-up and shared care following discharge from the Emergency Department for exacerbations of chronic disease. Can J Emerg Med. 2013; 13(Suppl 1):LOP05
- [Background] Hickey L, Hawton K, Fagg J, Weitzel H. Deliberate self-harm patients who leave the accident and emergency department without a psychiatric assessment: a neglected population at risk of suicide. J Psychosom Res. 2001 Feb;50(2):87-93. doi: 10.1016/s0022-3999(00)00225-7. PMID 11274665
- [Background] Suicide Prevention Resource Center. Caring for adult patients with suicide risk: A consensus guide for emergency departments [Internet]. Waltham (MA): Education Development Center Inc.; 2015 [cited 2017 Feb 20]. Available from: http://www.sprc.org/sites/default/files/EDGuide_full.pdf
- [Background] Suicide Prevention Resource Center. Preventing suicide among men in the middle years: Recommendations for suicide prevention programs [Internet]. Waltham (MA): Education Development Center Inc.; 2016 [cited 2017 Feb 20]. Available from: http://www.sprc.org/sites/default/files/resource-program/SPRC_MiMYReportFinal_0.pdf
- [Background] Allen NB. Cognitive therapy of depression. Aaron T Beck, A John Rush, Brian F Shaw, Gary Emery. New York: Guilford Press, 1979. Aust N Z J Psychiatry. 2002 Apr;36(2):275-8. doi: 10.1046/j.1440-1614.2002.t01-5-01015.x. No abstract available. PMID 11982561
- [Background] Hewitt PL, Flett GL, Weber C. Dimensions of perfectionism and suicide ideation. Cogn Ther Res. 1994; 18(5), 439-460.
- [Background] Kroenke K, Spitzer RL. The PHQ-9: A new depression diagnostic and severity measure. Psychiatr Ann. 2002; 32(9), 509-515.
- [Background] Prins A, Bovin MJ, Smolenski DJ, Marx BP, Kimerling R, Jenkins-Guarnieri MA, Kaloupek DG, Schnurr PP, Kaiser AP, Leyva YE, Tiet QQ. The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5): Development and Evaluation Within a Veteran Primary Care Sample. J Gen Intern Med. 2016 Oct;31(10):1206-11. doi: 10.1007/s11606-016-3703-5. Epub 2016 May 11. PMID 27170304
- [Background] Heisel MJ, Flett GL. Psychological resilience to suicide ideation among older adults. Clin Gerontol. 2008; 31(4), 439-640.
- [Background] Heisel MJ. Assessing experienced meaning in life among older adults: The development and initial validation of the EMIL. Int Psychogeriatr. 2009; 21 (Supplement 2), S172-S173.
- [Background] Mahalik JR, Locke BD, Ludlow LH, Diemer MA, Scott RP, Gottfried M, et al. Development of the conformity to masculine norms inventory. Psychol Men Masc. 2003; 4(1), 3-25.
- [Background] Brannon R, Juni S. A scale for measuring attitudes about masculinity. Psychological Documents. 1984; 14 (Doc.#2612).
- [Background] O'Neil JM, Helms BJ, Gable RK, David L, Wrightsman LS. Gender-role conflict scale: College men's fear of femininity. Sex Roles. 1986; 14(5), 335-350.
- [Background] D'Zurilla TJ, Nezu AM. Development and preliminary evaluation of the Social Problem-Solving Inventory. Psychol Assess. 1990; 2(2), 156-163.
- [Background] Hawton K, Williams K. Influences of the media on suicide. BMJ. 2002 Dec 14;325(7377):1374-5. doi: 10.1136/bmj.325.7377.1374. No abstract available. PMID 12480830
- [Background] Bisconer SW, Gross DM. Assessment of suicide risk in a psychiatric hospital. Prof Psychol Res Pr. 2007; 38(2), 143-149.
- [Background] Bethell J, Rhodes AE. Identifying deliberate self-harm in emergency department data. Health Rep. 2009 Jun;20(2):35-42. PMID 19728584
- [Background] Heisel, M. J., & Duberstein, P. R. (2016). Working sensitively and effectively to reduce suicide risk among older adults. (P. M. Kleespies, Ed.)The Oxford Handbook of Behavioural Emergencies and Crises (Vol. 1). Oxford University Press https://doi.org/10.1093/oxfordhb/9780199352722.013.25
- [Background] Health Canada. (2010). Acting on what we know: Preventing youth suicide in First Nations. Retrieved December 1, 2017, from http://www.hc-sc.gc.ca/fniah- spnia/pubs/promotion/_suicide/prev_youth-jeunes/index-eng.php#tphp.
- [Background] O'Connor E, Gaynes BN, Burda BU, Soh C, Whitlock EP. Screening for and treatment of suicide risk relevant to primary care: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 May 21;158(10):741-54. doi: 10.7326/0003-4819-158-10-201305210-00642. PMID 23609101
- [Background] Thompson, S. C., & Schlehofer, M. M. (2008). The many sides of control motivation: Motives for high, low, and illusory control. In J. Y. Shah & W. L. Gardner (Eds.), Handbook of motivation science. (pp. 41-56). New York, NY, US: The Guilford Press.
- [Background] Suicide Prevention Resource Center. (2015). Caring for adult patients with suicide risk: A consensus guide for emergency departments. Waltham, MA: Education Development Center, Inc.
- [Background] Clum, G. A., & Yang, B. (1995). Additional support for the reliability and validity of the Modified Scale for Suicide Ideation. Psychological Assessment, 7(1), 122-125. https://doi.org/10.1037/1040-3590.7.1.122.
- [Background] Kroenke, K., & Spitzer, R. L. (2002). The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals, 32(9), 509-515. https://doi.org/10.3928/0048- 5713-20020901-06.
- [Background] Wright JH, Wright AS, Albano AM, Basco MR, Goldsmith LJ, Raffield T, Otto MW. Computer-assisted cognitive therapy for depression: maintaining efficacy while reducing therapist time. Am J Psychiatry. 2005 Jun;162(6):1158-64. doi: 10.1176/appi.ajp.162.6.1158. PMID 15930065
- [Background] Hewitt, P. L., Flett, G. L., & Weber, C. (1994). Dimensions of perfectionism and suicide ideation. Cognitive Therapy and Research (Vol. 18). Retrieved from https://journals-scholarsportal-info.proxy.bib.uottawa.ca/pdf/00057967/v31i0002/229_dosiipi.xml.
- [Background] Arroll B, Goodyear-Smith F, Crengle S, Gunn J, Kerse N, Fishman T, Falloon K, Hatcher S. Validation of PHQ-2 and PHQ-9 to screen for major depression in the primary care population. Ann Fam Med. 2010 Jul-Aug;8(4):348-53. doi: 10.1370/afm.1139. PMID 20644190
- [Background] Heisel, M. J., & Flett, G. L. (2008). Psychological resilience to suicide ideation among older adults. Clinical Gerontologist, 31(4), 51-70. https://doi.org/10.1080/07317110801947177.
- [Background] Heisel, M. J. (2009). Assessing experienced meaning in life among older adults:The development and initial validation of the EMIL. International Psychogeriatrics, 21(S2), S172-173.
- [Background] Cocco, K. M., & Carey, K. B. (1998). Psychometric properties of the Drug Abuse Screening Test in psychiatric outpatients. Psychological Assessment, 10(4), 408-414. https://doi.org/10.1037/1040-3590.10.4.408.
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. https://doi.org/10.1207/s15327752jpa5201_2.
- [Background] Bouwmans C, De Jong K, Timman R, Zijlstra-Vlasveld M, Van der Feltz-Cornelis C, Tan Swan S, Hakkaart-van Roijen L. Feasibility, reliability and validity of a questionnaire on healthcare consumption and productivity loss in patients with a psychiatric disorder (TiC-P). BMC Health Serv Res. 2013 Jun 15;13:217. doi: 10.1186/1472-6963-13-217. PMID 23768141
- [Background] Niederkrotenthaler T, Fu KW, Yip PS, Fong DY, Stack S, Cheng Q, Pirkis J. Changes in suicide rates following media reports on celebrity suicide: a meta-analysis. J Epidemiol Community Health. 2012 Nov;66(11):1037-42. doi: 10.1136/jech-2011-200707. Epub 2012 Apr 21. PMID 22523342
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Derived] Hatcher S, Heisel MJ, Ayonrinde O, Corsi D, Edgar NE, Kennedy SH, Rizvi SJ, Schaffer A, Sinyor M. The BEACON study: an update to the protocol for a cohort study as part of an evaluation of the effectiveness of smartphone-assisted problem-solving therapy in men who present with intentional self-harm to emergency departments in Ontario. Trials. 2022 Oct 5;23(1):849. doi: 10.1186/s13063-022-06788-7. PMID 36199120
- [Derived] Hatcher S, Heisel M, Ayonrinde O, Campbell JK, Colman I, Corsi DJ, Edgar NE, Gillett L, Kennedy SH, Hunt SL, Links P, MacLean S, Mehta V, Mushquash C, Raimundo A, Rizvi SJ, Saskin R, Schaffer A, Sidahmed A, Sinyor M, Soares C, Taljaard M, Testa V, Thavorn K, Thiruganasambandamoorthy V, Vaillancourt C. The BEACON study: protocol for a cohort study as part of an evaluation of the effectiveness of smartphone-assisted problem-solving therapy in men who present with intentional self-harm to emergency departments in Ontario. Trials. 2020 Nov 13;21(1):925. doi: 10.1186/s13063-020-04424-w. PMID 33187542

DOCUMENTS (1):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT03473535/Prot_001.pdf